CLINICAL TRIAL: NCT04718454
Title: Retention and Wear Characteristic Assessment of OT Equator Smart Box Attachment Versus Ball Attachment for Mandibular Two Implant Assisted Over Denture , In-vitro Study
Brief Title: Retention and Wear Characteristic Assessment of OT Equator Smart Box Attachment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Amr Heshmat, lecturer od prosthodontic dep,, Cairo University
Other Study IDs: equator implant attachment
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Implant Breakage
Keywords: dental attachment; overdenture
MeSH Terms: interventions — Denture Precision Attachment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Equator attachment: Implant installation over epoxy resin model at the canine area on both sides following the surgical protocol of the implant placement,Equator Attachment fabrication is firmly screwed to the fixture on both sides at the canine region
  Interventions: Device: dental attachment
- ball attachment: Implant installation over epoxy resin model at the canine area on both sides following the surgical protocol of the implant placement,ball Attachment fabrication is firmly screwed to the fixture on both sides at the canine region
  Interventions: Device: dental attachment

INTERVENTIONS:
Device: dental attachment — This research aimed to evaluate the retentive power and wear of the smart box attachment use with tilted two implant assisted mandibular overdenture

SUMMARY:
This research aimed to evaluate the retentive power and wear of the smart box attachment use with tilted two implant assisted mandibular overdenture

DETAILED DESCRIPTION:
Implant supported overdenture can provide better mastication force than complete denture but less than the normal teeth . Most of the patient reported that implant supported overdenture has many superior features over the conventional complete denture in stability and retention Key factors related to successful treatment with overdentures include the number, location, and distribution of implants and choice of abutment. While the use of parallel implants that are widely distributed is generally desirable for optimal treatment, patients often present with challenging anatomical features, insufficient bone volume in all dimensions, and/or critical anatomy that precludes ideal placement of dental implants. Some clinicians may consider the ideal placement of implants for overdentures as parallel to each other and perpendicular to the occlusal plane of the denture Anatomical features associated with mandibular or maxillary edentulous ridges can range from straight or rounded to irregular and sharp ridges, and variability in bone width may limit potential implant sites for overdentures. Factors such as narrow bone volume, the inferior alveolar nerve being anterior or superior positioned, extensive bony undercuts, the inferior portion of the maxillary sinus, proximity to high-risk vascular structures, or a patient's desire to avoid additional surgical procedures may prompt a clinician to angulate a dental implant, which could result in the positioning of implants in non-ideal configurations.

Excessive angulation, increased maintenance and wear of inserts, and difficulty maintaining hygiene. Increased angulation may result in greater challenges to inserting and removing the prosthesis, which can become difficult for patients who are older and/or have limited dexterity. This challenge also can make it hard for patients to properly clean the inside of the retentive portion of the stud-style abutment and may increase wear of the retentive inserts Resilient Ball attachment most commonly used Ball attachment the simplest of all stud attachments which widely used because it is practical, effective, relatively low cost, less technique sensitive, ease of handling, minimal chair side time requirements and their possible applications with both root and implant-supported prostheses so it is used with non-splinted implants in clinical studies, it has been shown that changes in the retention of the prostheses occurred frequently. Both decrease and considerable increase in retention occurred as a result of attachment abrasion and micro movements during the mastication process The ball attachments showed only a few minor, easy manageable complications. Four out of 36 attachments gave reason for treatment. Two matrices loosened out of the mandibular denture and had to be fastened by adding acrylic resin after 1 and 4 weeks of loading. One patrix part of the ball attachment unsettled after 2 days of loading and was refastened. One ball attachment matrix lost its retention capacity and had to be reactivated after a period of 2 weeks. All these complications occurred in subjects where the implants were not perfectly parallel to each other positioned in the mandible. The loading conditions of these attachments were therefore not as favorable as for more parallel inserted implants A lack of parallelism of the implants creates considerable wear of the rubber rings in a relatively short time span.

Rhein 83, Italy, also has developed Smart Box, which could be used with the OT Equator in patients of extreme divergencies among the implants. The Smart Box has an inner tilting mechanism that enables a passive insertion with divergent implants up to 50 degrees(159).

ELIGIBILITY:
Inclusion Criteria:

* mandibular cast

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 10 mandibular edentolous casts
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Retention | 6 month
  Retention of OT equator smart box attachment versus ball attachment for mandibular two implant assisted over denture

SECONDARY OUTCOMES:
wear evaluation | 6 month
  wear evaluation of OT equator smart box attachment versus ball attachment for

REFERENCES:
- [Background] Ahmad R, Abu-Hassan MI, Chen J, Li Q, Swain MV. The Relationship of Mandibular Morphology with Residual Ridge Resorption Associated with Implant-Retained Overdentures. Int J Prosthodont. 2016 Nov/Dec;29(6):573-580. doi: 10.11607/ijp.4726. PMID 27824977